CLINICAL TRIAL: NCT03608319
Title: Phase 1, Open-Label, Randomized, 3-Way Crossover Relative Bioavailability of A4250 in Healthy Adult Subjects Under Fasting and Fed Conditions and When Sprinkled on Applesauce
Brief Title: Study of A4250 in Healthy Volunteers Under Fasting, Fed and Sprinkled Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Albireo (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A4250-004
Record Dates: First submitted 2018-07-13; First posted 2018-07-31 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: 3-Way Crossover Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single dose following overnight fast (Experimental)
  Interventions: Drug: A4250
- Single dose following high fat breakfast (Experimental)
  Interventions: Drug: A4250
- Single dose sprinkled on applesauce following overnight fast (Experimental)
  Interventions: Drug: A4250

INTERVENTIONS:
Drug: A4250 — 9.6 mg

SUMMARY:
The primary objective of this study is to determine the single-dose pharmacokinetics (PK) of A4250 when administered after a high-fat meal and when sprinkled on applesauce in healthy adult subjects.

DETAILED DESCRIPTION:
This is an open-label, randomized, 3-way crossover, food-effect and sprinkle study. On Day 1 of each period, subjects will receive a single oral dose of A4250 under 1 of 3 conditions: fasting, following a high-fat, high-calorie breakfast, or sprinkled on applesauce. Subjects will receive A4250 under each condition on one occasion. Blood samples for PK analysis will be collected for 18 hours following each study drug administration. There will be a washout period of at least 7 days between doses. Study participants will be contacted approximately 14 days after the last study drug administration to determine if any adverse event (AE) has occurred since the last study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male or female (of non-childbearing potential only), 19-55 years of age, inclusive, at screening.
2. Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dose and throughout the study as self-reported.
3. Body mass index (BMI) ≥ 18.0 and ≤ 28.0 kg/m2 at screening.
4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee at screening. Liver function (transaminases and serum bilirubin [total and direct]) must be within the upper limit of normal.
5. Female subjects must be of non-childbearing potential: i.e. must be post-menopausal or have undergone one of the following sterilization procedures at least 6 months prior to the first dose:

   * bilateral tubal ligation or bilateral salpingectomy;
   * hysterectomy;
   * bilateral oophorectomy;
6. A non-vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study drug.
7. If male, must agree not to donate sperm from the first dose until 90 days after the last dose.
8. Able to swallow multiple capsules.
9. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dose.
5. History or presence of hypersensitivity or idiosyncratic reaction to the study drug or related compounds.
6. History or presence of malabsorption syndrome (including clinically significant loose stool or diarrhea, as deemed by the PI) or cholestasis.
7. Female subjects with a positive pregnancy test or lactating.
8. Positive urine drug or alcohol results at screening or first check-in.
9. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
10. Unable to refrain from or anticipates the use of:

    • Any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements (including fiber supplements and laxatives) beginning 14 days prior to the first dose and throughout the study.
11. Is lactose intolerant.
12. Donation of blood or significant blood loss within 56 days prior to the first dose.
13. Plasma donation within 7 days prior to the first dose.
14. Participation in another clinical study within 30 days prior to the first dose. The 30-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2018-08-05 (Actual); Study Completion 2018-08-18 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of A4250 after a high fat meal | prior to dosing through 18 hours post dose
Area under the plasma concentration time curve from time zero extrapolated to infinity (AUC (0-inf)) of A4250 after a high fat meal | prior to dosing through 18 hours post dose
Area under the plasma concentration time curve from time zero to last measurable concentration (AUC(0-t)) of A4250 after a high fat meal | prior to dosing through 18 hours post dose
Maximum observed plasma concentration (Cmax) of A4250 sprinkled on applesauce | prior to dosing through 18 hours post dose
Area under the plasma concentration time curve from time zero extrapolated to infinity (AUC (0-inf)) of A4250 sprinkled on applesauce | prior to dosing through 18 hours post dose
Area under the plasma concentration time curve from time zero to last measurable concentration (AUC(0-t)) of A4250 sprinkled on applesauce | prior to dosing through 18 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No